CLINICAL TRIAL: NCT07312422
Title: An Open-label, Single-center, Single-arm Study to Evaluate the Efficacy and Safety of Low-dose Radiation Therapy Combined With Pultelimab and Standard Treatment in Patients With Advanced Pancreatic Cancer
Brief Title: LDRT Combined With Pucotenlimab and Standard Therapy for Advanced Pancreatic Cancer: A Single-Arm Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Yang, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pucotenlimab in PDAC
Record Dates: First submitted 2025-12-10; First posted 2025-12-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; PD-L1; PD-1 Inhibitor; LDRT; Proterizumab
Keywords: pancreatic cancer; PD-1 inhibitor; LDRT; immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT + Pucotenlimab + Chemotherapy (Experimental): Patients will receive low-dose radiotherapy (2Gy/1fx) on Day 1 of each cycle. On Day 2, patients will receive Pucotenlimab (200mg IV) combined with standard chemotherapy (investigator's choice of AG regimen or FOLFIRINOX regimen). Treatment cycles differ slightly based on the chemotherapy regimen chosen but are generally repeated every 3 weeks. Treatment continues until disease progression, unacceptable toxicity, or up to 2 years.
  Interventions: Radiation: Low-dose Radiotherapy; Biological: Pucotenlimab; Drug: AG regimen; Drug: FOLFIRINOX regimen

INTERVENTIONS:
Radiation: Low-dose Radiotherapy — Administered on Day 1 of each cycle. A single fraction of 2 Gy (2Gy/1fx) is delivered to the measurable tumor lesion using 3D-CRT or IMRT techniques.
Biological: Pucotenlimab — Administered intravenously (200 mg) on Day 2 of each cycle, every 3 weeks (q3w).
Drug: AG regimen — Gemcitabine (1000 mg/m^2) and Nab-paclitaxel (125 mg/m^2) administered intravenously on Day 1 and Day 8 of each 3-week cycle.
Drug: FOLFIRINOX regimen — Oxaliplatin (65 mg/m^2), Irinotecan (140 mg/m^2), Leucovorin (400 mg/m^2) on Day 1, followed by 5-FU (2400 mg/m^2) continuous infusion over 46 hours, every 3 weeks.

SUMMARY:
To investigate the activating effect of local lesion low-dose radiotherapy (2Gy) on the tumor immune microenvironment, and the efficacy, safety, and feasibility of its combination with pembrolizumab and standard therapy in patients with advanced pancreatic cancer. Concurrently, to preliminarily establish an efficacy prediction model for the early identification of patient populations who would benefit from the treatment, thereby providing a theoretical foundation for the implementation of precision medicine.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most malignant digestive tract tumors, with an extremely poor prognosis and a five-year survival rate of less than 10%. Its treatment options are limited. For patients with unresectable, advanced disease, systemic chemotherapy (such as the AG regimen or FOLFIRINOX regimen) is the standard treatment, but the efficacy remains unsatisfactory, with median overall survival struggling to exceed one year.

In recent years, immunotherapy represented by PD-1/PD-L1 inhibitors has achieved revolutionary success in various solid tumors (such as lung cancer, melanoma), bringing hope for long-term survival to patients with advanced cancer. However, in the field of pancreatic cancer, immunotherapy monotherapy has repeatedly faced setbacks. Multiple clinical studies show that immune checkpoint inhibitors have a very low response rate (typically <5%) in unselected patients with advanced pancreatic cancer, with the vast majority failing to benefit. This characteristic of being an immunologically "cold" tumor is largely attributed to the unique tumor microenvironment (TME) of pancreatic cancer: a highly fibrotic stroma, minimal infiltration of cytotoxic T lymphocytes (CTLs), and an abundance of immunosuppressive cells (such as regulatory T cells (Tregs), myeloid-derived suppressor cells (MDSCs)). These factors collectively create a state of immune exclusion and immunosuppression, preventing immune cells from recognizing and attacking tumor cells.

To convert "cold tumors" into "hot tumors," researchers are actively exploring various combination strategies. Among them, the combination of radiotherapy (RT) and immunotherapy shows great potential. Traditionally, radiotherapy was considered merely a local treatment modality. However, recent studies have found that it also has the abscopal effect - where irradiation of one lesion can lead to the shrinkage of non-irradiated, distant lesions. This suggests that radiotherapy can activate a systemic anti-tumor immune response. It is noteworthy that low-dose radiotherapy (e.g., 2Gy) plays a unique role in this process. Unlike high-dose radiotherapy, which primarily causes DNA double-strand breaks in tumor cells, low-dose radiotherapy is more capable of inducing immunogenic cell death (ICD), prompting tumor cells to release antigens and danger signal molecules, thereby enhancing antigen presentation by dendritic cells (DCs) and initiating a T-cell immune response. Multiple preclinical studies have confirmed that 2Gy radiotherapy can effectively promote the cross-presentation of tumor-specific antigens, reduce immunosuppression in the microenvironment, and increase the infiltration of lymphocytes into the tumor site, creating favorable conditions for immunotherapy to take effect.

Based on the above evidence, we propose the following scientific hypothesis: For patients with advanced pancreatic cancer who are insensitive to immunotherapy monotherapy, preemptive intervention using low-dose radiotherapy is expected to remodel the tumor immune microenvironment (TIME), converting it from "cold" to "hot." Subsequently, the follow-up combination of a PD-1 inhibitor (Pucotenlimab) and standard chemotherapy could not only activate the immune system via radiotherapy but also further kill tumor cells and expose more tumor antigens through chemotherapy, potentially suppressing immunosuppressive cells. The synergistic effect of these three modalities is expected to achieve a "1+1+1>3" outcome, potentially breaking through the current therapeutic bottleneck for advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of gender;
* ECOG score of 0 to 1;
* Patients with histologically or cytologically confirmed pancreatic malignancy;
* No prior treatment with PD-1 or PD-L1 inhibitors;
* Presence of a radiotherapeutically eligible target lesion (excluding bone metastases);
* Subjects voluntarily participate in the study and provide signed informed consent.

Exclusion Criteria:

* Previous history of radiotherapy;
* Uncontrolled chronic infectious or non-infectious diseases, including but not limited to: medication-refractory heart failure, poorly controlled hypertension, etc.;
* Active or clinically uncontrolled severe infections;
* History of psychoactive drug abuse that cannot be abstained from, or patients with psychiatric disorders;
* Pregnant or lactating women, or patients of childbearing potential who are unwilling or unable to adopt effective contraceptive measures;
* Other conditions deemed by the investigator as potentially affecting the conduct of the clinical study or the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 weeks
  Overall objective tumor response rate

SECONDARY OUTCOMES:
DCR | 2 years
  Disease control rate
PFS | 2 years
  Progression free Survial

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No